CLINICAL TRIAL: NCT04301466
Title: Efficacy and Safety of Qi Zhi Tong Luo Capsule in Vascular Cognitive Impairment: a Randomized, Double-blind, Placebo- Controlled, Multicentre Study
Brief Title: Efficacy and Safety of Qi Zhi Tong Luo Capsule in Vascular Cognitive Impairment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Shanxi Zhendong Pharmacy Co., Ltd (Industry)
Responsible Party: Principal Investigator, Jinzhou Tian, Vice president, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B20020126
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Vascular Cognitive Impairment; Qi Zhi Tong Luo Capsule; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qi Zhi Tong Luo group (Experimental): Patients were receiveed Qi Zhi Tong Luo Capsule 4 capsules, 2 times per day for 24 weeks. Each capsule was weighted 0.5g. Qi Zhi Tong Luo capsule (batch number: 20140805) were produced by Shanxi Zhendong Pharmaceutical Co., Ltd.
  Interventions: Drug: Qi Zhi Tong Luo capsule
- Placebo group (Placebo Comparator): Patients were allocated to placebo, 4 capsules, 2 times per day for 24 weeks. Placebo (batch number: 20140805) were produced by Shanxi Zhendong Pharmaceutical Co., Ltd.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Qi Zhi Tong Luo capsule — Patients were receiveed Qi Zhi Tong Luo Capsule 4 capsules, 2 times per day for 24 weeks. QZTL capsule, a traditional Chinese medicine. Each capsule was weighted 0.5g.
  Arms: Qi Zhi Tong Luo group
Drug: Placebos — Patients were allocated to placebo, 4 capsules, 2 times per day for 24 weeks.To preserve blinding, the placebo had an identical taste and appearance to the experimental drugs. Placebo (batch number: 20140805) were produced by Shanxi Zhendong Pharmaceutical Co., Ltd.
  Arms: Placebo group

SUMMARY:
Qi Zhi Tong Luo (QZTL) capsule, a traditional Chinese herbal medicine, which was used to treat stoke-related symptoms, include trouble speaking, paralysis and trouble walking. This study aimed to evaluate the efficacy and safety of QZTL capsule in the treatment of vascular cognitive impairment. This study was designed as randomized, double-blind, parallel, placebo-controlled, multicentre trial. It consisted of a single-blind run-in period using placebo only (2 weeks) and a double-blind treatment phase after randomization (24 weeks), and follow-up 12 weeks after withdrawal.The primary efficacy variables included changes from baseline in the Clinical Dementia Rating scale-Sum Box (CDR-SB) and the Mini-mental State Examination (MMSE) after 24 weeks of treatment. The secondary efficacy measurements include the Clock Drawing Test (CDT), Hopkins Verbal Learning Test (HVLT) and Ability of Daily Living (ADL).

ELIGIBILITY:
Inclusion Criteria:

1. Decline in cognitive function from a prior baseline and impairment in at least 1 cognitive domain, the domain of cognition including executive function(Trail Making Test-part A(Chinese version,150s)>98s)), memory function decline (Hopkins verbal learning test free recall(36 points) <18.5 points), language function decline (Boston naming test (Chinese version 30 items)<22 points), and visuo-spatial functions (Clock drawing test(10 points)<8.5 points) ;
2. Evidence of cerebrovascular disease relies on structural magnetic resonance imaging (MRI) , history and clinical feature. The neuroimaging should include at least one of following: a) a single large vessel infarction which was sufficient to cause cognition decline; b) infarction at a single strategic place was sufficient to cause severe cognition decline( the thalamus, angular gyrus, and basal ganglia, including the caudate nucleus and globus pallidus); c) multiple lacunar infarctions (≥3) outside the brainstem, or 2 lacunar infarcts at key locations, a single lacunar focus with extensive white matter lesions(WMLs) ; d) extensive and integrated WMLs(Fazekas scale≥3 points) ; e) intracranial hemorrhage in key parts, or ≥2 intracranial hemorrhages; f) combination of above.
3. There was a clear temporal relationship between a vascular event and onset of cognitive deficit, cognitive impairment should appear within 3 months after a stroke, or abrupt deterioration, or stepwise progression of deficits; or cognitive impairment may be related to vascular factors, the Hachinski Ischemia scale (HIS) score ≥7;
4. And the patients must have adequate vision and hearing to participate in study assessments;
5. Have a stable caregiver;
6. Can read simple articles and write simple sentences;
7. Informed consent, signed informed consent by legal guardian.

Exclusion Criteria:

1. Evidence of other reasons caused cognitive impairment, like Alzheimer disease, frontotemporal dementia, Parkinson disease dementia, dementia with Lewy bodies, Huntington disease, etc;
2. Subdural hematoma, traffic hydrocephalus, brain tumor, thyroid disease, vitamin deficiency, or other diseases which can lead to cognitive impairment;
3. Major depression (Hamilton depression rating scale [HAMD] ≥17) or other mental disorders ;
4. History of drug or alcohol abuse in the past 6 month;
5. History of epilepsy;
6. Patients with myasthenia gravis;
7. Subject cannot complete related test due to severe neurologic deficits;
8. Other uncontrolled chronic illnesses, like severe cardiovascular disease (severe arrhythmia, myocardial infarction within 3 months, severe heart failure(New York Heart Association Functional Classification III and IV,); uncontrolled hypertension, diabetes);
9. Severe liver or kidney dysfunction (alanine aminotransferase or aspartate transaminase was more than 1.5 times the upper limit of normal, or serum creatinine was more than the upper limit of normal);
10. Concomitant use of the anticonvulsants, antipsychotics, cholinomimetic drugs, anticholinergic agents, anti-Parkinson drugs, cholinesterase inhibitors, memantine, nootropic drug, nimodipine, anticholinergic or anticholinergic antidepressant or anxiolytic and other cognition enhancers within 1 month;
11. Severe asthma and chronic obstructive pulmonary disease;
12. Patients with severe indigestion, gastrointestinal obstruction, gastric or duodenal ulcers;
13. Patients with glaucoma;
14. History of hypersensitivity to the treatment drugs;
15. Participate in other clinical study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Changes of Clinical Dementia Rating-Sum of the Boxes scale (CDR-SB) from baseline | week 0, 12, 24,36
  CDR-SB is a standard for disease grading in clinical studies of dementia and is used for overall endpoint assessment in clinical trials. The CDR-SB scores from 0-18 points, and a higher score indicates higher impairment.
Changes of Mini-mental State Examination(MMSE from baseline | week 0, 12, 24,36
  MMSE, 0-30 points, a lower score means severe global cognition impairment, which is used for overall endpoint assessment in clinical trials.

SECONDARY OUTCOMES:
Changes of Hopkins Verbal Learning Test from baseline | week 0, 12, 24,36
  0-48 points, higher score indicates better memory function
Changes of Clock drawing test from baseline | week 0, 12, 24,36
  0-10 points, with higher scores indicating better visuo-spatial function
Changes of Ability of daily living scale from baseline | week 0, 12, 24,36
  0-56 points, higher score means severe ability daily living function

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital ,Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China